CLINICAL TRIAL: NCT02853786
Title: Influence of Language Environment in Children With Cochlear Implants
Brief Title: Language Environment in Children With Cochlear Implants
Acronym: ISLODA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9678; 2016-A00155-46 (Other: ANSM)
Record Dates: First submitted 2016-07-07; First posted 2016-08-03 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Language Development
Keywords: cochlear implant; language environment; speech therapy assessment; LENA technology
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LENA and advices (Experimental): With the LENA results, we will advise the parents how to improve the language environment to help their children with CIs for their language development
  Interventions: Behavioral: LENA and advice
- LENA without advices (Active Comparator): Regular speech therapy follow blindly the results of LENA
  Interventions: Other: LENA without advice

INTERVENTIONS:
Behavioral: LENA and advice — Language recording with the LENA device, with the LENA results, we will advise the parents how to improve the language environment to help their children with CIs for their language development
  Arms: LENA and advices
Other: LENA without advice — Language recording with the LENA device. Regular speech therapy follow blindly the results of LENA
  Arms: LENA without advices

SUMMARY:
The Language Environment Analysis (LENA) system is a specific tool for the language environment analysis. Children aged from 18 months to 6 years old, with cochlear implants (CIs), wear an electronic device during a day and their language interactions are registered. Then the investigators can analyze with a specific software four different parameters (adult words, conversational turns, child vocalizations and media exposure) and compare them to the language ability of the children assessed by a speech therapist. With the results, the speech therapist can advise the parents how to improve the language environment to help their children with CIs for their language development. Parents are encouraged to follow these advices at home during few months (5 months +/-1 month). Then there is a new registration of the LENA device and another language assessment are performed, to see if there is any improvement. The investigators also measure the family participation.

Hypothesis : There is an influence of the language environment measured by the LENA system on language development in children with cochlear implants.

DETAILED DESCRIPTION:
Over 24 months the investigators will recruit 90 patients with cochlear implants (CIs) in 2 centers.

Each patient will follow during 5 months and will have three or five visits according to the arm.

ELIGIBILITY:
Eligibility Criteria:*

Inclusion criteria:

* Congenital profound deaf children
* aged from 18 months to 5 years old 11 months
* with a cochlear implant at least since 6 months
* regular following in speech therapy

Exclusion criteria:

* non-francophone parents
* syndrome (like CHARGE syndrome) or aplasia
* partial insertion of the electrode array
* associated troubles (Autism Spectrum Disorders, mental retardation…)
* visual troubles
* irregular use of the cochlear implant (externe part)
* absence of parental consent

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Change in language environment measured by LENA system | At the inclusion, and 5 months after the inclusion

SECONDARY OUTCOMES:
Change in language ability measured by the Grammatical Analysis Of Elicited Language Presentence level (GAEL-P) | At the inclusion, and 5 months after the inclusion
Change in language ability measured by a vocabulary scale with peabody images (EVIP) (EVIP) | At the inclusion, and 5 months after the inclusion

IPD SHARING:
Plan to Share IPD: No